CLINICAL TRIAL: NCT01020383
Title: A Phase 2 Randomized, Open Label Clinical Trial in High Risk Percutaneous Coronary Intervention (PCI) Patients Receiving Standard Antithrombotic Treatment Plus Either ALX-0081 or GPIIb/IIIa Inhibitor (ReoPro®) Over a Period of 24 Hours
Brief Title: Comparative Study of ALX-0081 Versus GPIIb/IIIa Inhibitor in High Risk Percutaneous Coronary Intervention (PCI) Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ablynx, a Sanofi company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALX-0081-2.1/09
Record Dates: First submitted 2009-11-23; First posted 2009-11-24 (Estimated); Last update posted 2023-04-04 (Actual); Status verified 2019-01

CONDITIONS: Unstable Angina; Non ST Segment Elevation Myocardial Infarction (NSTEMI); Stable Angina (Associated With High Risk PCI)
MeSH Terms: conditions — Angina, Unstable; Non-ST Elevated Myocardial Infarction; Angina, Stable | interventions — caplacizumab; Abciximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ALX-0081 (Experimental)
  Interventions: Drug: ALX-0081
- GPIIb/IIIa inhibitor (Active Comparator)
  Interventions: Drug: ReoPro®

INTERVENTIONS:
Drug: ALX-0081 — 4 i.v. bolus injections, once every 6 hours; first dose of 6 mg, three subsequent doses of 4 mg
  Arms: ALX-0081
Drug: ReoPro® — 0.25 mg/kg i.v. bolus injection followed by continuous i.v. infusion of 0.125 µg/kg/min (to a max. of 10 µg/min) for 12 hours
  Arms: GPIIb/IIIa inhibitor

SUMMARY:
This is a multicenter, randomized and open-label Phase II study to compare the safety, tolerability and biological effectiveness of ALX-0081 versus the GPIIb/IIIa inhibitor ReoPro® in high risk PCI patients.

Patients will receive standard treatment with acetylsalicylic acid (ASA) plus clopidogrel and heparin. Eligible patients will be randomly assigned to receive open-label study treatment with either ALX-0081 or ReoPro®. Patients will be stratified according to PCI type (elective or ad-hoc) and stent type (bare metal stent or drug eluting stent).

ELIGIBILITY:
Inclusion Criteria:

* Have unstable angina or NSTEMI,or stable angina with at least 2 factors indicating a high risk PCI as follows: patient related: diabetic patients, renal failure (glomerular filtration rate < 60), reduced left ventricular ejection fraction < 35%, age > 75 years, female gender and/or lesion/anatomy related: SYNTAX score > 26, bifurcation lesions, multi-vessel disease, intracoronary thrombus.
* Adequate hematological function including platelets > 100000/mm3.
* Body mass index (BMI) ≥18 kg/m2 and ≤ 35 kg/m2.
* Aged ≥ 18 years old.
* Women of childbearing potential must be practicing a medically acceptable contraceptive regimen. Only males who do not want to father children during the study and in the first 4 months after treatment may be included in the study. During this period, safe contraception is mandatory. Male patients who are sexually active must use a condom during intercourse and ensure that the female partner uses a reliable contraceptive method, or they must refrain from sexual intercourse during the first 4 months after treatment.
* Patients must be accessible for follow-up.
* Have a sufficient command to read and understand all instructions necessary for giving informed consent and participating in the study.
* Have signed and dated written informed consent prior to any study-related procedures.

Exclusion Criteria:

* Previous (within 30 days) treatment with GPIIb/IIIa inhibitors (such as ReoPro®).
* ST-elevation myocardial infarction (STEMI).
* Chronic total occlusion of a coronary artery.
* Scheduled rotablator procedure.
* PCI of the arterial or venous by-pass graft.
* Any contra-indication for ReoPro®.
* Major organ dysfunction, infection or any serious underlying medical condition that would impair the ability of the patient to receive protocol treatment.
* Known hypersensitivity to human/humanized antibodies.
* Women who are pregnant or lactating.
* Dementia or significantly altered mental status that would prohibit understanding the study procedures and giving informed consent.
* Use of vitamin K antagonists and/or Factor Xa inhibitors within 4 weeks prior to admission to the Hospital Intensive Care Unit.
* Use of GPIIa/IIIb inhibitors other than ReoPro®; prasugrel, bivalirudin and fondaparinux prior to and throughout the study.
* Known history of acquired or congenital bleeding disorder, coagulopathy or platelet disorder.
* Evidence of active pathological bleeding at screening or history of clinically significant bleeding (such as gastrointestinal or genitourinary) within the last 6 months prior to screening visit, unless the cause has been definitely corrected
* History of intracranial bleeding (e.g. hemorrhagic stroke, subdural hematoma, subarachnoid hemorrhage) or history of hemorrhagic retinopathy.
* History of ischemic stroke or TIA, within the past year prior to screening or known structural cerebral vascular lesion (e.g. arteriovenous malformation, aneurysm).
* History of New York Heart Association class III or IV congestive heart failure or history of severe, uncontrolled cardiac arrhythmias at screening.
* Planned elective surgical operation or major invasive procedures or traumas from 30 days prior to screening to completion of the study at Day 30 (the decision of what constitutes a major invasive procedure or trauma will be at the discretion of the investigator in conjunction with review and approval by the Medical Monitor).
* Use of another investigational drug or device within previous 30 days (12 weeks for investigational devices, e.g. unapproved stents) prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 364 (Actual)
Dates: Start 2009-09; Primary Completion 2011-04 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of bleeding classified by the following criteria: TIMI major bleeding events, TIMI minor bleeding events, bleeding events requiring medical attention, defined as TIMI minimal bleeding events | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Josefin-Beate Holz, MD, Study Director — Ablynx NV
Locations (39):
- Austria (3):
  - Graz
  - Linz
  - Vienna
- Belgium (6):
  - Aalst
  - Charleroi
  - Genk
  - Jette
  - Liège
  - Yvoir
- Czechia (3):
  - Brno
  - Prague
  - Ústí nad Labem
- Germany (7):
  - Bad Nauheim
  - Coburg
  - Dortmund
  - Hamburg
  - Limburg
  - Oldenburg
  - Rostock
- Israel (5):
  - Ashkelion
  - Haifa
  - Jerusalem
  - Rehovot
  - Tel Litwinsky
- Poland (13):
  - Bielsko-Biala
  - Dąbrowa Górnicza
  - Gdynia
  - Grodzisk Mazowiecki
  - Katowice
  - Kędzierzyn
  - Kościerzyna
  - Krakow
  - Lódz
  - Poznan
  - Torun
  - Warsaw
  - Wroclaw
- Switzerland (2):
  - Lausanne
  - Lugano

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org